CLINICAL TRIAL: NCT00143923
Title: Heart Strategies Concentrating On Risk Evaluation (Heart SCORE) Study
Brief Title: Novel Strategies for Reducing Heart Disease Risk Disparities
Acronym: HeartSCORE
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Responsible Party: Principal Investigator, Steven E. Reis, MD, Professor of Medicine, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: STUDY20060247; PA DOH ME-02-384 (Other Grant/Funding Number: Commonwealth of Pennsylvania)
Record Dates: First submitted 2005-09-01; First posted 2005-09-02 (Estimated); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Cardiovascular Diseases
Keywords: Cardiovascular Diseases; Risk Factors; Sleep disordered breathing; Environmental exposures; Cognitive Function
MeSH Terms: conditions — Cardiovascular Diseases; Sleep Apnea Syndromes | interventions — Nutritional Status; Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- 1 (Active Comparator): Intervention: 6 months of individualized advice regarding Nutrition, Exercise, Stress Management Counseling for participants who are at intermediate or high Framingham risk for CVD and are randomized to Arm 1
  Interventions: Behavioral: Nutrition, Exercise, Stress Management Counseling
- 2 (Placebo Comparator): Intervenition: 6 months of Usual care for participants who are at intermediate or high Framingham risk for CVD and are randomized to Arm 2. No active Nutrition, Exercise, Stress Management Counseling
  Interventions: Other: usual care
- 3 (No Intervention): No intervention for all participants who are at low Framingham risk for CVD or have preexisting CVD prior to study entry/ No active Nutrition, Exercise, Stress Management Counseling

INTERVENTIONS:
Behavioral: Nutrition, Exercise, Stress Management Counseling — Individualized advice
  Arms: 1
Other: usual care — usual care
  Arms: 2

SUMMARY:
This Western Pennsylvania-based study will (1) improve cardiovascular risk stratification to identify high-risk populations, (2) identify differences in cardiovascular risk, (3) evaluate mechanisms for population differences in cardiovascular risk, and (4) implement a multidisciplinary community-based intervention program to decrease cardiovascular risk in high-risk populations.

This is a prospective cohort study of 2,000 residents of the state of Pennsylvania. All participants will undergo assessments of traditional and nontraditional risk factors to identify and determine the mechanisms of population disparities in cardiovascular risk. 800 participants who are at intermediate or high risk of cardiovascular disease will be randomly assigned to either (1) usual care/"advice only"; or (2) a multidisciplinary behavioral modification program to determine the most effective approach to reduce or eliminate differences in cardiovascular risk among high risk populations. All participants will undergo long-term follow-up for cardiovascular events.

DETAILED DESCRIPTION:
Well-established disparities exist in the prevalence and outcome of cardiovascular disease related to race and socioeconomic status (SES). Our previous work confirms these disparities and suggests that they may be related to population differences in the prevalence of nontraditional cardiovascular risk factors. We propose that these disparities can be significantly reduced or eliminated by (1) a community-based intervention program that incorporates a multidisciplinary education program led by a behavioral interventionalist, a nutritionist and an exercise physiologist, and (2) a novel approach to cardiovascular risk stratification that considers population differences in traditional and nontraditional risk factors and subclinical atherosclerosis.

To successfully implement this program, particularly in traditionally underserved communities, we have formalized a partnership between the University of Pittsburgh School of Medicine and Graduate School of Public Health, the Pittsburgh Mind-Body Center, and the Pittsburgh Theological Seminary, Urban League of Pittsburgh, and Jewish Healthcare Foundation. This partnership is positioned to study the following specific aims:

1. To determine whether a community-based intervention program that incorporates a multidisciplinary education program led by a behavioral interventionalist, a nutritionist, and an exercise physiologist can reduce racial and socioeconomic disparities in cardiovascular risk in intermediate and high risk populations.
2. To ascertain whether a comprehensive assessment of nontraditional risk factors and subclinical atherosclerosis can provide incremental value above and beyond traditional risk assessment in identifying individuals at high cardiovascular risk.

ELIGIBILITY:
Inclusion Criteria:

* Men and women age 45-75 years

Exclusion Criteria:

* Comorbidity that is expected to limit life expectancy to <5 years
* Inability to undergo baseline or annual follow-up visits
* Pregnancy (exclude women from Xray studies)

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2000 (Actual)
Dates: Start 2003-03; Primary Completion 2029-12 (Estimated); Study Completion 2029-12 (Estimated)

PRIMARY OUTCOMES:
CVD Events | 20 years
  Major adverse cardiovascular events

CONTACTS AND LOCATIONS:
Overall Officials: Steven E Reis, MD, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No